CLINICAL TRIAL: NCT05769920
Title: A Phase 1 Dose-Escalation Study Evaluating the Safety, Tolerability, and Pharmacokinetics of TTHX1114(NM141) Ophthalmic Solution In Healthy Adult Volunteers
Brief Title: Dose Escalation TTHX1114 Ophthalmic Solution
Acronym: EPI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trefoil Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: NM141-001
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Corneal Epithelial Degeneration
MeSH Terms: interventions — Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TTHX1114 Dose Level 1 (Experimental): TTHX1114(NM141) Ophthalmic Solution (DL1): 1 drop (gtt) to the Study Eye (SE) twice daily for a total of 7 days
  Interventions: Drug: TTHX1114(NM141) Ophthalmic Solution
- TTHX1114 Dose Level 2 (Experimental): TTHX1114(NM141) Ophthalmic Solution (DL2): 1 drop (gtt) to the Study Eye (SE) twice daily for a total of 7 days
  Interventions: Drug: TTHX1114(NM141) Ophthalmic Solution
- TTHX1114 Dose Level 3 (Experimental): TTHX1114(NM141) Ophthalmic Solution (DL3): 1 drop (gtt) to the Study Eye (SE) twice daily for a total of 7 days
  Interventions: Drug: TTHX1114(NM141) Ophthalmic Solution
- TTHX1114 Dose Level 4 (Experimental): TTHX1114(NM141) Ophthalmic Solution (DL4): 1 drop (gtt) to the Study Eye (SE) twice daily for a total of 7 days
  Interventions: Drug: TTHX1114(NM141) Ophthalmic Solution

INTERVENTIONS:
Drug: TTHX1114(NM141) Ophthalmic Solution — Eye drop twice daily

SUMMARY:
Dose escalation 3+3 design with accelerated titration 4 dose levels

DETAILED DESCRIPTION:
This is a 28-day open-label dose-escalation study. TTHX1114(NM141) Ophthalmic Solution: 1 drop (gtt) to the Study Eye (SE) twice daily for a total of 7 days. Four planed dose levels, accelerated titration DL1 and DL2, standard 3+3 design.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18 to 65 years of age, Female subjects of child-bearing potential must be non-pregnant
* Able to provide voluntary written informed consent
* Normal ocular function (BCVA 20/20) and anatomy
* Available for and agree to all study procedures including inpatient monitoring, follow-up visits, sample collection, study treatment administration
* Body mass index 18.5 to 35 kg/m^2
* Demonstrated ability to self-administer eye drops

Exclusion Criteria:

* Clinically significant co-morbid ocular conditions
* Co-morbid medical conditions requiring treatment
* Active ocular infection within the 2 weeks prior to Day 1
* Active non-ocular infection requiring antibiotics within the 2 weeks prior to Day 1
* Use of systemic or dermatological cytotoxic chemotherapy within the 1 month prior to Day 1
* Planned contact lens use during the study period
* Use of any investigational product within the 1 month prior to Day 1
* Corticosteroid use in the 1 month prior to Day 1
* Major surgery within the 3 months prior to Day 1
* History of dependence on alcohol or drugs of abuse
* History of intolerance, hypersensitivity, or significant allergy to any drug compound, food, or other substance
* Any other reason (e.g., serious systemic disease or uncontrolled medical condition) that, in the opinion of the Investigator could increase the subject's risk, interfere with the interpretation of the study results, or affect the subject's ability to provide informed consent or comply with the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 28 days
  Important Medical Events (ocular) related to study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tremblay, Study Director — Trefoil Therapeutics.com
Locations (1):
- Trefoil Clinical Site #132, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No